CLINICAL TRIAL: NCT04085484
Title: Effects of Two Different Parenteral Nutrition Regimes on Nutrient Intakes, Growth and Plasma Electrolytes in Very Low Birth Weight Infants
Acronym: PUMPA
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Magnus Domellöf, Professor, Principal Investigator, Umeå University
Other Study IDs: 2011/417-31M
Record Dates: First submitted 2019-09-03; First posted 2019-09-11 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Nutrition Disorder, Infant
Keywords: preterm
MeSH Terms: conditions — Infant Nutrition Disorders; Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants born between 1 Feb 2010 and 18 Feb 2012: Infants born between 1 February 2010 and 18 February 2012, before the concentrated PN regime was implemented (Original PN group: n = 81).
- Infants born between 19 Feb 2012 and 30 Sep 2013: Infants born between 19 February 2012 and 30 September 2013, after the concentrated PN regime was implemented (Concentrated PN group: n = 53).
  Interventions: Dietary Supplement: More concentrated parenteral nutrition solution

INTERVENTIONS:
Dietary Supplement: More concentrated parenteral nutrition solution — This study is a single-center retrospective observational study comparing two cohorts of very low birth weight (VLBW, birth weight < 1500 grams) infants who received parenteral nutrition (PN) either before or after a concentrated PN regime was implemented into clinical use. Both PN regimes were based on standardized PN solutions.
  Groups: Infants born between 19 Feb 2012 and 30 Sep 2013

SUMMARY:
A single-center retrospective observational study comparing two cohorts of very low birth weight (VLBW, birth weight < 1500 grams) infants who received parenteral nutrition (PN) either before or after a concentrated PN regime was implemented into clinical use. Primary outcome is weight SDS at 28 days.

DETAILED DESCRIPTION:
This study is a single-center retrospective observational study comparing two cohorts of very low birth weight (VLBW, birth weight < 1500 grams) infants who received parenteral nutrition (PN) either before or after a concentrated PN regime was implemented into clinical use. Both PN regimes were based on standardized PN solutions with the possibility to complement with additive nutritional products according to individual assessment by the attending physician. To meet recommended macronutrient intakes, in 2012 a concentrated parenteral nutrition regime was implemented into clinical use at the neonatal intensive care unit in Umeå University hospital, Sweden. However, there is a lack of data on how changes in nutrient intakes affect growth and electrolyte status in preterm infants. Recent studies have demonstrated an increased incidence of hypokalaemia, hypophosphatemia and hypercalcaemia in infants who received enhanced parenteral energy and protein intakes.

This study is a single-center retrospective observational study comparing two cohorts of very low birth weight (VLBW, birth weight < 1500 grams) infants who received parenteral nutrition (PN) either before or after a concentrated PN regime was implemented into clinical use. Both PN regimes were based on standardized PN solutions with the possibility to complement with additive nutritional products according to individual assessment by the attending physician.

ELIGIBILITY:
Inclusion Criteria:

* All infants VLBW infants admitted to the neonatal intensive care unit at Umeå University Hospital, Sweden, within 24 hours after birth and treated there for ≥ 7 days, during 1 February 2010 and 30 September 2013.

The infants were divided into two groups:

1. infants born between 1 February 2010 and 18 February 2012, before the concentrated PN regime was implemented (Original PN group: n = 81), and
2. infants born between 19 February 2012 and 30 September 2013, after the concentrated PN regime was implemented (Concentrated PN group: n = 53).

Exclusion Criteria:

* Infants with chromosomal or severe congenital anomalies known to affect nutritional intakes and / or growth were excluded from the analyses.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants VLBW infants admitted to the neonatal intensive care unit at Umeå University Hospital, Sweden, within 24 hours after birth and treated there for ≥ 7 days, during 1 February 2010 and 30 September 2013.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Weight | 28 days
  Primary outcome is weight Standard Deviation Score (SDS)

SECONDARY OUTCOMES:
Length and head circumference | First 28 days of life
  Length (SDS score) and head circumference (SDS score) Nutritional intakes: All enteral and parenteral intakes during the first 28 postnatal days.
  Health outcome: Neonatal morbidities (including respiratory dristress syndrome (RDS), bronchopulmonary dysplasia (BPD), necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP), interaventricular hemorrhage (IVH) mm.) Nutritional biomarkers: Daily measurements of plasma sodium, potassium, calcium and phosphate during the first postnatal week.
Nutrient intakes (macronutrients and electrolytes) | First 28 days of life
  Energy intake (kcal/kg), protein intake (g/kg), fat (g/kg), carbohydrates (g/kg), sodium (mg/kg), potassium (mg/kg), calcium (mg/kg), phosphorous (mg/kg)
Biomarkers of nutrition (electrolytes and glucose) | First 28 days of life
  plasma sodium (mmol/L), potassium (mmol/L), calcium (mmol/L), phosphate (mmol/L), glucose (mmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spath C, Sjostrom ES, Domellof M. Higher Parenteral Electrolyte Intakes in Preterm Infants During First Week of Life: Effects on Electrolyte Imbalances. J Pediatr Gastroenterol Nutr. 2022 Sep 1;75(3):e53-e59. doi: 10.1097/MPG.0000000000003532. Epub 2022 Jun 20. PMID 35726971